CLINICAL TRIAL: NCT01335919
Title: Non-invasive Continuous Hemoglobin in Pediatric Medicine: a Comparison Between Standard of Care CBC Hemoglobin (ADVIA 2120®) and the New Masimo® SpHb® Neonatal Sensor
Brief Title: Neonatal Non-Invasive Hemoglobin Determination
Status: Withdrawn | Type: Observational
Why Stopped: Company is redesigning measuring tool.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-007757
Record Dates: First submitted 2011-02-02; First posted 2011-04-15 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Surgical Procedures; Infant, Newborn; Infant, Low Birth Weight
Keywords: Hemoglobin; Monitoring, Physiologic; Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonate: Subjects admitted for surgery or to the pediatric intensive care unit (PICU) or neonatal intensive care unit (NICU) who require daily and/or multiple blood samples for hemoglobin measurement.

SUMMARY:
The purpose of this study is to evaluate hemoglobin (Hgb) measurement by Masimo-developed pulse co-oximetry in pediatric patients weighing less than 3 kilograms (Kg).

DETAILED DESCRIPTION:
This collaborative study with Masimo Corporation will involve 2 phases. In the first phase of this study, 25 subjects weighing 0.5 to 3.0 kg will be recruited and hemoglobin values will be obtained from the non-invasive probe at the same time as blood samples are routinely drawn for Hgb analysis using the cyanomethemoglobin method (ADVIA 2121). Masimo Corporation will use this data to calibrate or modify the hemoglobin reading (SpHb®) sensors and monitors. All results and conclusions from this phase will be discussed with the investigation team in order to determine if additional subjects are needed (at increments of 25 subjects at a time). Once the sensor designs have been optimized, another group of patients will be studied to document the accuracy and precision of the hemoglobin reading (SpHb®) measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females weighing 0.5 kg to 3 kg.
2. Neonates and infants and children admitted to the Children's Hospital of Philadelphia (CHOP)operating room (OR), PICU and NICU where hemoglobin measurements are anticipated.
3. Parental/guardian permission (informed consent)

Exclusion Criteria:

1. Subjects where blood samples are obtained through access types other than venous or arterial (e.g: intraosseous).
2. Subject weighing more than 3 kg.
3. Subjects who are too small or with any anatomical limitations that would preclude proper attachment of the adhesive sensor.
4. Any skin rash on the intended site of measurement. Severe allergy to adhesive tapes.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted for a surgical procedure or admitted to the PICU or NICU where hemoglobin determinations are expected.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Non-invasive, photoplethysmographic, hemoglobin reading (SpHb®) | up to 5 minutes
  The primary endpoint is comparing at least one simultaneous non-invasive, photoplethysmographic, hemoglobin reading (SpHb®) and one invasive hemoglobin measurements (Hb) for each subject. (SpHb® vs. Hb)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Jablonka, MD, Principal Investigator — Children's Hospital of Philadelphia